CLINICAL TRIAL: NCT02508077
Title: A Prospective Study of FOLFIRI Plus Panitumumab in Extended RAS Wild Type and BRAF Wild Type Metastatic Colorectal Cancer With Acquired Resistance to Prior Cetuximab (or Panitumumab) Plus Irinotecan-Based Therapy and Who Failed at Least One Subsequent Non-anti-EGFR Containing Regimen
Brief Title: FOLFIRI and Panitumumab in Treating Patients With RAS and BRAF Wild-Type Metastatic Colorectal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor Accrual
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15117; NCI-2015-01241 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 118713; 15117 (Other: City of Hope Comprehensive Cancer Center)
Record Dates: First submitted 2015-07-22; First posted 2015-07-24 (Estimated); Results first posted 2018-08-16 (Actual); Last update posted 2018-08-16 (Actual); Status verified 2018-07

CONDITIONS: Recurrent Colorectal Carcinoma; Stage IVA Colorectal Cancer; Stage IVB Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Fluorouracil; dehydroftorafur; Irinotecan; Leucovorin; Panitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (panitumumab and FOLFIRI) (Experimental): Patients receive panitumumab IV over 30-90 minutes, irinotecan hydrochloride IV over 90 minutes, leucovorin calcium PO, and fluorouracil IV over 46 hours on day 1. Courses repeat every 2 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Fluorouracil; Drug: Irinotecan Hydrochloride; Other: Laboratory Biomarker Analysis; Drug: Leucovorin Calcium; Biological: Panitumumab

INTERVENTIONS:
Drug: Fluorouracil — Given IV
  Other Names: 5-Fluoro-2,4(1H, 3H)-pyrimidinedione; 5-Fluorouracil; 5-Fluracil; 5-FU; AccuSite; Actino-Hermal; Adrucil; Arumel; Cytosafe; Efudex; Efurix; Fiverocil; Fluoro Uracil; Fluoroplex; Fluouracil; Flurablastin; Fluracedyl; Fluracil; Fluril; Fluroblastin; Flurox; Ribofluor; Ro 2-9757; Ro-2-9757; Timazin
Drug: Irinotecan Hydrochloride — Given IV
  Other Names: Campto; Camptosar; Camptothecin 11; Camptothecin-11; CPT 11; CPT-11; U-101440E
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Leucovorin Calcium — Given PO
  Other Names: Adinepar; Calcifolin; Calcium (6S)-Folinate; Calcium Folinate; Calcium Leucovorin; Calfolex; Calinat; Cehafolin; Citofolin; Citrec; Citrovorum Factor; Cromatonbic Folinico; Dalisol; Disintox; Divical; Ecofol; Emovis; Factor, Citrovorum; Flynoken A; Folaren; Folaxin; FOLI-cell; Foliben; Folidan; Folidar; Folinac; Folinate Calcium; folinic acid; Folinic Acid Calcium Salt Pentahydrate; Folinoral; Folinvit; Foliplus; Folix; Imo; Lederfolat; Lederfolin; Leucosar; leucovorin; Rescufolin; Rescuvolin; Tonofolin; Wellcovorin
Biological: Panitumumab — Given IV
  Other Names: ABX-EGF; ABX-EGF Monoclonal Antibody; ABX-EGF, Clone E7.6.3; MoAb ABX-EGF; Monoclonal Antibody ABX-EGF; Vectibix

SUMMARY:
This phase II trial studies how well fluorouracil, leucovorin calcium, and irinotecan hydrochloride (FOLFIRI) together with panitumumab work in treating patients with colorectal cancer that expresses the RAS and B-Raf proto-oncogene, serine/threonine kinase (BRAF) wild-type genes, has spread from the original site of growth to another part of the body (metastatic), resists the effects of treatment with prior cetuximab (or panitumumab) plus irinotecan hydrochloride-based therapy, and who have failed at least one subsequent non-anti-epidermal growth factor receptor (EGFR) containing treatment regimen. Drugs used in chemotherapy, such as fluorouracil, leucovorin calcium, and irinotecan hydrochloride, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving more than one drug (combination chemotherapy) may kill more tumor cells. Monoclonal antibodies, such as panitumumab, may block tumor growth in different ways by targeting certain cells. Giving FOLFIRI together with panitumumab may be an effective treatment for colorectal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Estimate the response rate (RR) and progression-free survival (PFS) with FOLFIRI + panitumumab in patients with acquired resistance to panitumumab (or cetuximab) + irinotecan (irinotecan hydrochloride)-based therapy after a documented clinical response or prolonged PFS and following progression on a subsequent non-anti-EGFR containing regimen in extended RAS wild-type and BRAF wild-type patients.

SECONDARY OBJECTIVES:

I. Estimate the overall survival (OS) in the re-challenge populations.

II. Describe the safety of re-challenge in this population.

III. Investigate the impact of PFS, RR on prior anti-EGFR + irinotecan-based exposure on the response and PFS on the current study.

TERTIARY OBJECTIVES:

I. Collect serial plasma samples to investigate the incidence of RAS and BRAF mutation in circulating free deoxyribonucleic acid (DNA) at baseline, every 2 months, and at the time to progression (and following progression when feasible).

II. Collect serial plasma samples for future biomarker exploration, including the potential investigation of micro-ribonucleic acid (RNA).

OUTLINE:

Patients receive panitumumab intravenously (IV) over 30-90 minutes, irinotecan hydrochloride IV over 90 minutes, leucovorin calcium orally (PO), and fluorouracil IV over 46 hours on day 1. Courses repeat every 2 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then every 3 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have the ability to understand and the willingness to sign a written informed consent document
* Participant must be willing to comply with study and/or follow-up procedures
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Life expectancy of 3 >= months
* Histologically confirmed colon or rectal cancer with metastatic disease
* Extended RAS and BRAF wild type status documented on archival tumor tissue or on fresh biopsy if no archival tissue present
* Measurable disease defined by at least 1 lesion >= 1 cm
* Documented objective response or stable disease lasting for 6 months or more to last prior anti-EGFR (cetuximab or panitumumab) in combination with irinotecan or FOLFIRI
* Progression within 6 weeks following their last dose of anti-EGFR therapy
* Treatment with a non-EGFR targeting regimen following progression on anti-EGFR plus irinotecan-based therapy
* At least 4 months from prior anti-EGFR therapy prior to start of study treatment
* At least three weeks from any non-anti-EGFR therapy prior to start of study treatment; any number of prior therapies is permitted
* Adequate recovery in the investigators opinion from any clinically significant toxicity from prior therapy
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L
* Hemoglobin (Hgb) >= 9 g/dL without transfusions
* Platelets (PLT) >= 100 x 10^9/L without transfusions
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) and/or alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x upper limit of normal (ULN); patient with liver metastases =< 5 x ULN
* Total bilirubin =< ULN
* Creatinine =< 1.5 mg/dL
* Magnesium >= 1.2mg/dL or 0.5 mmol/L
* Negative serum beta-human chorionic gonadotropin (HCG) test (female patient of childbearing potential only), to be performed locally within the screening period
* Agreement by females of childbearing potential and sexually active males to use an effective method of contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for three months following duration of study participation; should a woman become pregnant or suspect that she is pregnant while participating on the trial, she should inform her treating physician immediately

Exclusion Criteria:

* History of severe anti-EGFR toxicity requiring drug discontinuation or dose-modification within the first 4 months of prior anti-EGFR therapy
* History of intolerance to irinotecan at dose-intensity of 125 mg/m^2/2 weeks or lower
* History of intolerance to 5-FU at dose-intensity of 1800 mg/m^2/2 weeks or lower
* Current use (or planned use during the treatment period) of other investigational agents, or biological, chemotherapy, radiation or other anti-tumor therapy
* Co-medication that may interfere with study results; e.g. immuno-suppressive agents other than corticosteroids, such as systemic cyclosporine and tacrolimus
* No St John's wort supplement or other herbal supplementation is allowed while on trial; patients are not to take grapefruit juice during study treatment
* Use of drugs known to inhibit UDP glycosyltransferase 1 family, polypeptide A1 gene (UGT1A1), such as Atazanavir, Gemfibrozil, Indinavir, or Ketoconazole while on study treatment; (patients using these drugs must not take these drugs on the day study treatment begins and for the duration of study treatment)
* Planned use of strong cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4) inhibitors or CYP3A4 inducers while on study treatment unless deemed clinically necessary with no reasonable alternatives and with expressed permission from the principal investigator
* If on anticoagulation, participant must be on stable therapeutic dose prior to enrollment
* Impairment of gastrointestinal function or gastrointestinal disease (e.g., active ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, extensive small bowel resection)
* Major surgery =< 3 weeks prior to starting study drug or who have not recovered from side effects of such procedure
* Unstable pulmonary embolism, deep vein thrombosis, or other significant arterial/venous thromboembolic event =< 30 days before enrollment
* Clinically significant cardiovascular disease (including myocardial infarction, unstable angina, symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia) =< 6 months prior to enrollment
* History of interstitial lung disease (ILD) eg, interstitial pneumonitis, pulmonary fibrosis or evidence of ILD on baseline chest computed tomography (CT) or magnetic resonance imaging (MRI)
* Other active malignancies except cervical carcinomas in situ or clinically insignificant non-melanoma skin cancers
* Clinically significant uncontrolled illness or active infections
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to irinotecan, 5-FU, leucovorin or any of the products to be administered during dosing
* Pregnant women and women who are lactating; breastfeeding should be discontinued if the mother is enrolled on this study
* Any other condition that would, in the Investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns or compliance with clinical study procedures, e.g., infection/inflammation, intestinal obstruction, unable to swallow medication, social/psychological issues, etc
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-02-16 (Actual); Primary Completion 2017-09-13 (Actual); Study Completion 2017-09-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marwan Fakih, Principal Investigator — City of Hope Comprehensive Cancer Center
Locations (4):
- United States (4):
  - City of Hope Medical Center, Duarte, California
  - City of Hope Antelope Valley, Lancaster, California
  - City of Hope Rancho Cucamonga, Rancho Cucamonga, California
  - South Pasadena Cancer Center, South Pasadena, California

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Panitumumab and FOLFIRI): Patients receive 6mg/kg panitumumab IV over 30-90 minutes, 180mg/m2 irinotecan hydrochloride IV over 90 minutes, 400mg/m2 leucovorin calcium PO, and 2400mg/m2 fluorouracil IV over 46 hours on day 1. Courses repeat every 2 weeks in the absence of disease progression or unacceptable toxicity.
  Fluorouracil: Given IV
  Irinotecan Hydrochloride: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Leucovorin Calcium: Given PO
  Panitumumab: Given IV
Period: Overall Study
Arm/Group | Treatment (Panitumumab and FOLFIRI)
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Panitumumab and FOLFIRI)
Number analyzed (Participants) | 1
Age, Continuous [Median (Full Range); unit: years] | 57 [57 to 57]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: 4-month Progression-free Survival (PFS) Rate
Description: PFS is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first. Will be estimated using the product-limit method of Kaplan and Meier. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum on study (including baseline sum), or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: At 4 months
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (Panitumumab and FOLFIRI)
Number analyzed (Participants) | 1
percentage of participants | 0

ADVERSE EVENTS:
Time Frame: Adverse events occurred over a period of 12 weeks.
Description: "Other Adverse Events" include all events that were not severe adverse events regardless of grade or relation to treatment.
Arm/Group | Treatment (Panitumumab and FOLFIRI)
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Panitumumab and FOLFIRI) (N=1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
blood anion gap decreased. (Blood and lymphatic system disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (2)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Study was terminated early due to poor accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-07): https://cdn.clinicaltrials.gov/large-docs/77/NCT02508077/Prot_SAP_000.pdf